CLINICAL TRIAL: NCT04594967
Title: The Community for Successful Ageing (ComSA) Patient-Centered Care (COPACC) Study: Utilization, Health and Economic Evaluation of a Community-Based Primary Care Geriatric Hub at Whampoa, Singapore.
Brief Title: The COPACC Study: Utilization, Health and Economic Evaluation of a Community-Based Primary Care Geriatric Hub at Whampoa
Status: Completed | Type: Observational
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Tsao Foundation (Unknown); National Healthcare Group, Singapore (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017/00352
Record Dates: First submitted 2020-10-06; First posted 2020-10-20 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2020-10

CONDITIONS: Delivery of Health Care; Health Services; Costs and Cost Analysis; Quality of Life
Keywords: patient-centred care; patient-centred medical home; older adults; complex needs; healthcare utilisation; economic evaluation; cost analysis; health services research

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient-centred care home (PCMH) — New model of care defined by care provision by a team of people centered in the community that is both proactive and coordinated to improve the health and wellness of the people in that community.

SUMMARY:
This study evaluates the Community for Successful Ageing (ComSA) Patient-Centered Medical Home (PCMH), a model of community-based primary care geriatric hub at Whampoa, Singapore.

DETAILED DESCRIPTION:
This study evaluates the Community for Successful Ageing (ComSA) Patient-Centered Medical Home (PCMH), a model of community-based primary care geriatric hub at Whampoa, Singapore. This study aims to evaluate the impact of ComSA PCMH on health service utilisation, healthcare cost, clinical quality and effectiveness, as well as patient activation, quality of life, satisfaction and experience of care. The first component of the study is a single arm prospective pre-post cohort design, which aims to evaluate the impact on enrolled patients' self-reported health outcomes, experience of care, and cost effectiveness. The second component of the study evaluates the quality of the implementation processes via clinical quality indicators. The third component is a match-controlled retrospective pre-post study design, which aims to evaluate the impact on healthcare utilisation. Data sources include both survey data and administrative data.

ELIGIBILITY:
Key inclusion criteria:

i. Aged 40 years and above ii. Lives in Whampoa, Singapore iii. Enrolled in PCMH after 1 September 2017

Exclusion criteria:

i. Aged less than 40 years ii. Does not live in Whampoa Singapore

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Older adults aged 40 years and above who reside in Whampoa, Singapore, and have complex healthcare needs.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Healthcare utilisation: Primary care | Change from baseline to post-3 months, and to post-6 months
  Primary care visits
Healthcare utilisation: Inpatient visits | Change from baseline to post-3 months, and to post-6 months
  Inpatient visits
Healthcare utilisation: Specialist outpatient care | Change from baseline to post-3 months, and to post-6 months
  Specialist outpatient clinic visits
Healthcare utilisation: A&E | Change from baseline to post-3 months, and to post-6 months
  A&E visits
Patient-reported outcome measure for patient activation | Change from baseline to post-3 months, and to post-6 months
  PAM-13
Patient-reported outcome measure for quality of life | Change from baseline to post-3 months, and to post-6 months
  EQ-5D-5L
Patient-reported outcome measure for quality of life in old age | Change from baseline to post-3 months, and to post-6 months
  CASP-19
Patient experience of care | 6 months
  CAHPS
Economic evaluation and cost analysis | Change from baseline to post-3 months, and to post-6 months
  Cost comparison between intervention group and non-intervention group

CONTACTS AND LOCATIONS:
Overall Officials: Chek Hooi Wong, Principal Investigator — Geriatric Education and Research Institute
Locations (1):
- Geriatric Education and Research Institute, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim ZZB, Mohamed Kadir M, Ginting ML, Vrijhoef HJM, Yoong J, Wong CH. Early Implementation of a Patient-Centered Medical Home in Singapore: A Qualitative Study Using Theory on Diffusion of Innovations. Int J Environ Res Public Health. 2021 Oct 24;18(21):11160. doi: 10.3390/ijerph182111160. PMID 34769680